CLINICAL TRIAL: NCT01246830
Title: The Use of 2D and 3D Imaging Modalities and Its Influence on Diagnosis and Treatment Planning in Orthodontics
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S52731
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2010-09

CONDITIONS: Orthodontics; Malocclusion; Impacted Tooth; Cephalometry; Cone-Beam Computed Tomography; Panoramic Radiography
MeSH Terms: conditions — Malocclusion; Tooth, Impacted | interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3D cephalometric analysis
  Interventions: Radiation: Cone-beam computed tomography (CBCT)
- 2D cephalometric analysis
  Interventions: Radiation: Panoramic radiograph, Cephalometric radiograph

INTERVENTIONS:
Radiation: Panoramic radiograph, Cephalometric radiograph — 2D images that are used for orthodontic treatment planning
  Groups: 2D cephalometric analysis
Radiation: Cone-beam computed tomography (CBCT) — CBCT data will be used in 3D cephalometric analysis softwares
  Groups: 3D cephalometric analysis

SUMMARY:
Research questions:

1. Will the panoramic images derived from cone beam CT data give better diagnostic ability than conventional panoramic radiographs?
2. Will 3D cephalometric analysis offer the orthodontists and surgeons better information for treatment planning?
3. Will the 3D cephalometric analysis give more accurate treatment plan and better treatment outcome?

General hypothesis and special aims

Overall aims:

* To compare 2D versus 3D cephalometric analysis: treatment planning and therapeutic outcome.
* To determine the accuracy and diagnostic ability and usability of the 3D cephalometric analysis.
* To evaluate the diagnostic ability and usability of the panoramic image derived from cone beam CT data as compared to 2D panoramic images.
* To evaluate the value of the cone beam CT data in cephalometric analysing process for orthodontic and maxillofacial surgery treatment.

Hypotheses:

1. The availability of the 3D cephalometric analysis influences the orthodontic and maxillofacial treatment plan and decision, and might change the treatment outcome.
2. Panoramic images derived from cone beam CT data may provide equal information for diagnosis as conventional panoramic images.
3. Cone beam CT will be able to replace "classic orthodontic imaging" being more time and dose efficient and having a beneficial effect on treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* age 12-25 years old
* Patients with malocclusions
* Patients with jaw relation defect both with or without the need of orthognathic surgery
* Patients with maxillofacial defects: tumors and trauma
* Patients with eruption problems: embedded or impacted teeth which have to be removed

Exclusion Criteria:

* Patients with congenital deformities
* Patients with systemic diseases that may effect the growth formation: growth factor defect and thyroid hormone defect.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are seeking orthodontic and maxillofacial surgery treatments at the University Hospital Leuven with the need of conventional panoramic radiographs, cephalometric radiographs and cone beam CT images.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cephalometric analysis | at treatment planning step and after 2 years of treatment
  linear and angular cephalometric measurement

SECONDARY OUTCOMES:
outcome of orthodontic treatment | after 2 years of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Katholieke Universiteit Leuven, Leuven
  - University Hospital Leuven, Leuven

REFERENCES:
- [Background] Broadbent BH. A new x-ray technique and its application to orthodontia. Angle Orthodontist 1931;51: 115-150
- [Background] Swennen GR, Schutyser F, Barth EL, De Groeve P, De Mey A. A new method of 3-D cephalometry Part I: the anatomic Cartesian 3-D reference system. J Craniofac Surg. 2006 Mar;17(2):314-25. doi: 10.1097/00001665-200603000-00019. PMID 16633181
- [Background] Swennen GR, Schutyser F. Three-dimensional cephalometry: spiral multi-slice vs cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2006 Sep;130(3):410-6. doi: 10.1016/j.ajodo.2005.11.035. PMID 16979502
- [Background] Olszewski R, Cosnard G, Macq B, Mahy P, Reychler H. 3D CT-based cephalometric analysis: 3D cephalometric theoretical concept and software. Neuroradiology. 2006 Nov;48(11):853-62. doi: 10.1007/s00234-006-0140-x. Epub 2006 Sep 29. PMID 17009024
- [Background] Scarfe WC, Farman AG. What is cone-beam CT and how does it work? Dent Clin North Am. 2008 Oct;52(4):707-30, v. doi: 10.1016/j.cden.2008.05.005. PMID 18805225
- [Background] Carter L, Farman AG, Geist J, Scarfe WC, Angelopoulos C, Nair MK, Hildebolt CF, Tyndall D, Shrout M; American Academy of Oral and Maxillofacial Radiology. American Academy of Oral and Maxillofacial Radiology executive opinion statement on performing and interpreting diagnostic cone beam computed tomography. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Oct;106(4):561-2. doi: 10.1016/j.tripleo.2008.07.007. No abstract available. PMID 18928899
- [Background] Hassan B, van der Stelt P, Sanderink G. Accuracy of three-dimensional measurements obtained from cone beam computed tomography surface-rendered images for cephalometric analysis: influence of patient scanning position. Eur J Orthod. 2009 Apr;31(2):129-34. doi: 10.1093/ejo/cjn088. Epub 2008 Dec 23. PMID 19106265
- [Background] Lou L, Lagravere MO, Compton S, Major PW, Flores-Mir C. Accuracy of measurements and reliability of landmark identification with computed tomography (CT) techniques in the maxillofacial area: a systematic review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Sep;104(3):402-11. doi: 10.1016/j.tripleo.2006.07.015. Epub 2006 Oct 27. PMID 17709072
- [Background] de Oliveira AE, Cevidanes LH, Phillips C, Motta A, Burke B, Tyndall D. Observer reliability of three-dimensional cephalometric landmark identification on cone-beam computerized tomography. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Feb;107(2):256-65. doi: 10.1016/j.tripleo.2008.05.039. Epub 2008 Aug 20. PMID 18718796
- [Background] Periago DR, Scarfe WC, Moshiri M, Scheetz JP, Silveira AM, Farman AG. Linear accuracy and reliability of cone beam CT derived 3-dimensional images constructed using an orthodontic volumetric rendering program. Angle Orthod. 2008 May;78(3):387-95. doi: 10.2319/122106-52.1. PMID 18416632
- [Background] Brown AA, Scarfe WC, Scheetz JP, Silveira AM, Farman AG. Linear accuracy of cone beam CT derived 3D images. Angle Orthod. 2009 Jan;79(1):150-7. doi: 10.2319/122407-599.1. PMID 19123719
- [Background] Olszewski R, Tanesy O, Cosnard G, Zech F, Reychler H. Reproducibility of osseous landmarks used for computed tomography based three-dimensional cephalometric analyses. J Craniomaxillofac Surg. 2010 Apr;38(3):214-21. doi: 10.1016/j.jcms.2009.05.005. Epub 2009 Jul 1. PMID 19574058
- [Background] Proffit WR, Fields HW Jr., Sarver DM. Contemporary Orthodontics. 4th ed, Mosby Inc., Elsevier Science, Philadelphia, 2006.
- [Background] White SC, Pharoah MJ. The evolution and application of dental maxillofacial imaging modalities. Dent Clin North Am. 2008 Oct;52(4):689-705, v. doi: 10.1016/j.cden.2008.05.006. PMID 18805224